CLINICAL TRIAL: NCT05340361
Title: In vivO Study of assessmeNt for Efficacy and safetY of Zotarolimus-eluting Stent OVERexpansion With Optical Coherence Tomography (ONYSOVER Trial)
Brief Title: Efficacy and Safety of Zotarolimus-eluting Stent Overexpansion With OCT
Acronym: ONYSOVER
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Severance Hospital (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Yongcheol Kim, Clinical Associate Professor, Yonsei University
Other Study IDs: 9-2021-0176
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Optical Coherence Tomography; Stent
Keywords: coronary artery disease; optical coherence tomography; stenting
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- In vivo: OCT examination is performed using a frequency-domain OCT system (C7 DragonflyTM OPTISTM Imaging Catheter, Abbott Vascular, Santa Clara, CA, USA) with a 5.4 or 7.5 cm total pullback length according to a non-occlusive technique. The procedure is performed via radial or femoral access with a ≥6 Fr guiding catheter. The OCT catheter is advanced over the 0.014-inch PCI wire and the implanted stent was crossed after administration of intracoronary nitrates of 200 µg. For blood clearing, contrast media was injected through the guiding catheter with an automated power injector. The standard infusion rate was 4 mL/s for 4 seconds with 250 PSI. Follow-up OCT image acquisition was achieved with the same method. After post-PCI OCT, we evaluate the factor regarding post-PCI optimization target by European Expert Consensus.
  Interventions: Device: Optical coherence tomography-guided percutaneous coronary intervention; Device: Optical coherence tomography-guided Onyx family stent expansion

INTERVENTIONS:
Device: Optical coherence tomography-guided percutaneous coronary intervention — OCT examination is performed using a frequency-domain OCT system (C7 Dragonfly OPTIS Imaging Catheter, Abbott Vascular, Santa Clara, CA, USA) with a 5.4 or 7.5 cm total pullback length according to a non-occlusive technique. The procedure is performed via radial or femoral access with a ≥6 Fr guiding catheter. The OCT catheter is advanced over the 0.014-inch PCI wire and the implanted stent was crossed after administration of intracoronary nitrates of 200 µg. For blood clearing, contrast media was injected through the guiding catheter with an automated power injector. The standard infusion rate was 4 mL/s for 4 seconds with 250 PSI. Follow-up OCT image acquisition was achieved with the same method. After post-PCI OCT, we evaluate the factor regarding post-PCI optimization target by European Expert Consensus.
  Other Names: Zotarolimus-eluting stent (Onyx family stent, Medtronic, Santa Rosa, CA, USA)
Device: Optical coherence tomography-guided Onyx family stent expansion — 1. Expansion of 2.25, 3.0, and 4.0 mm Onyx family stent@ nominal pressure
  2. OCT pullback
  3. Expansion with over 0.5mm sized non-compliant balloon of each stent
  4. OCT pullback
  5. Expansion with over 1.0mm sized non-compliant balloon of each stent
  6. OCT pullback
  7. Expansion with over 1.25~1.5mm sized non-compliant balloon of each stent
  8. OCT pullback
  9. Evaluation of polymer status with overexpansion assessed by an electric microscope

SUMMARY:
Investigators aimed to evaluate efficacy and safety of expansion capacity of zotarolimus-eluting Stent assessed by optical coherence tomography (OCT) in vivo study.

DETAILED DESCRIPTION:
Single stent implantation (also called "provisional stenting") is currently the preferred technique for percutaneous coronary interventions on the majority of unprotected left main (LM) or non-LM bifurcations. During provisional stenting, proximal optimization technique (POT), proved to correct both the proximal main vessel (MV) malapposition and/or optimize the side branch (SB) ostium strut opening for proper wire re-crossing into the distal cell, might be crucial step and may warrant improved long-term clinical outcomes in the setting of major proximal and distal reference vessel size mismatch (like often in LM bifurcation or diffuse tapered long lesion).

Recently, second-generation drug-eluting stent (DES) implantation is recommended over BMS for PCI in patients with ischemic heart disease (IHD) due to superior efficacy and safety. However, percutaneous coronary intervention (PCI) with DES for lesion with the discrepancy of proximal and distal reference vessel size, such as LM or non-LM bifurcation lesion, diffuse tapered long lesion, and ectatic or aneurysmal coronary artery, is challenging due to stent optimization because expert consensus recommend that stent diameter is selected by distal reference diameter, which need stent overexpansion for POT.

OCT is a utility that can accurately measure reference vessel diameter and lesion length pre-PCI, which is useful for stent optimization by a suitable stent selection and pre- and post-interventional strategies. OCT also demonstrated higher sensitivity to detect stent malapposition, edge dissection, and tissue prolapsed than IVUS post-PCI. Thus, OCT-guided PCI can be helpful to optimize DES implantation in patients with dilated coronary arteries despite the potential limitation of depth penetration and attenuation images by thrombus.

Zotarolimus-eluting stent (Onyx family stent, Medtronic, Santa Rosa, CA, USA) was developed in response to the demand for stents with improved radiographic visibility. It has a novel thin strut composite wire stent platform that is covered with the same zotarolimus-eluting durable polymer coating as its predecessors. The metallic stent platform consists of a composite wire made from a dense platinum-iridium core, which makes the struts radiopaque, and an outer layer of cobalt-chromium alloy. The dense core also allows for reduced strut thickness, which might be associated with a decreased risk of stent thrombosis.

Onyx family stent has been labeled for maximum stent inner diameter by easy crowns platform (2.00-2.5 mm, 6.5 Crowns; 2.75-3.0 mm, 8.5 crowns; 3.5-4.0 mm, 9.5 crowns; 4.5-5.0 mm; 10.5 crowns). However, safety and efficacy of DES overexpansion is still concerned as safety of efficacy of there are limited data regarding Onyx family stent overexpansion in vivo.

This study aims to evaluate the safety and efficacy of Onyx family stent overexpansion for lesion with the discrepancy between proximal and distal reference vessel which need stent overexpansion for POT, assessed by OCT, providing high-resolution (10 µm) imaging which enables the detection of strut fracture, malapposition.

ELIGIBILITY:
Inclusion Criteria:

* Patients, ≥19 years of age, who were diagnosed with IHD requiring stent implantation for lesion with size discrepancy between proximal and distal reference diameter over 1mm, such as tapered long lesion or bifurcation lesion, confirmed by OCT
* The decision to participate voluntarily in this study and the written consent of the patient

Exclusion Criteria:

* Patients with hypersensitivity or contraindication to antiplatelet treatment
* Female of childbearing potential, who possibly plans to become pregnant any time after enrollment into this study.
* Patients with a life expectancy shorter than 1 year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IHD had a discrepancy between proximal and distal reference vessels requiring stent implantation and considering stent overexpansion will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal stent overexpansion (%) | Through procedure completion, up to 24 hours
  defines as the ratio of the maximal stent diameter to each diameter of stent

SECONDARY OUTCOMES:
Stent strut fracture | Through procedure completion, up to 24 hours
  defines as none or fewer visible stent strut on the cross-sectional view by performing OCT within stented segments (In in vivo and in vitro groups)
Absolute average stent diameter (mm) in the maximal stent expansion site | Through procedure completion, up to 24 hours
  Absolute average stent diameter (mm) in the maximal stent expansion site ((In in vivo and in vitro groups)
Grade of polymer damage assessed by electron microscope | Through procedure completion, up to 1-month
  Grade of polymer damage assessed by electron microscope (In in vitro group)

CONTACTS AND LOCATIONS:
Locations (1):
- Yongin Severance Hospital, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
I'll share the IPD if other researchers have good reason.